CLINICAL TRIAL: NCT00506415
Title: A 48-Week, Multicenter, Randomized, Double-Blind, Parallel-Group Evaluation of the Comparative Efficacy, Safety, and Tolerability of Exelon® 10 and 15 cm^2 Patch in Patients With Mild to Moderate Alzheimer's Disease (AD) Showing Functional and Cognitive Decline
Brief Title: Comparative Efficacy, Safety, and Tolerability of Rivastigmine 10 and 15 cm^2 Patch in Patients With Alzheimer's Disease (AD) Showing Cognitive Decline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CENA713D2340
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's; Patch; Cognitive; Decline
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Open label: Rivastigmine (5 cm^2 / 10 cm^2) (Experimental): Rivastigmine 5 cm^2 transdermal patch once a day during the first 4 weeks of open label treatment followed by rivastigmine 10 cm^2 transdermal patch once a day from week 4 to week 24, 36 or 48.
  Interventions: Drug: Rivastigmine 5 cm^2; Drug: Rivastigmine 10 cm^2
- Double blind: Rivastigmine (10 cm^2) (Experimental): Rivastigmine transdermal patch 10 cm^2 and placebo to rivastigmine 15 cm^2 once daily for 48 weeks during the double blind period.
  Interventions: Drug: Rivastigmine 10 cm^2; Drug: Placebo to 15 cm^2 patch
- Double blind: Rivastigmine (15 cm^2) (Experimental): Rivastigmine transdermal patch 15 cm^2 and placebo to rivastigmine 10 cm^2 once daily for 48 weeks during double blind period.
  Interventions: Drug: Rivastigmine 15 cm^2; Drug: Placebo to 10 cm^2 patch
- Extended open label Rivastigmine (10 cm^2) (Experimental): Rivastigmine 10 cm^2 transdermal patch once a day during 48 weeks open label treatment running in parallel to the double blind period.
  Interventions: Drug: Rivastigmine 10 cm^2

INTERVENTIONS:
Drug: Rivastigmine 5 cm^2 — 5 cm^2 transdermal patch
  Other Names: Exelon®
  Arms: Open label: Rivastigmine (5 cm^2 / 10 cm^2)
Drug: Rivastigmine 10 cm^2 — 10 cm^2 transdermal patch.
  Other Names: Exelon®
  Arms: Double blind: Rivastigmine (10 cm^2); Extended open label Rivastigmine (10 cm^2); Open label: Rivastigmine (5 cm^2 / 10 cm^2)
Drug: Rivastigmine 15 cm^2 — 15 cm^2 transdermal patch.
  Other Names: Exelon®
  Arms: Double blind: Rivastigmine (15 cm^2)
Drug: Placebo to 15 cm^2 patch — Placebo of rivastigmine transdermal patch 15 cm^2.
  Arms: Double blind: Rivastigmine (10 cm^2)
Drug: Placebo to 10 cm^2 patch — Placebo of rivastigmine transdermal patch 10 cm^2.
  Arms: Double blind: Rivastigmine (15 cm^2)

SUMMARY:
The purpose of this study was to support the optimal use of rivastigmine patch in long-term treatment of Alzheimer's Disease in patients demonstrating functional and cognitive decline at the target maintenance dose of rivastigmine patch 10 cm^2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 50 and 85 years of age with a diagnosis of probable Alzheimers Disease,
* Baseline Mini-Mental State Examination (MMSE) score 10-24 inclusive,
* A primary caregiver willing to accept responsibility for supervising treatment, assessing the patient's condition throughout the study, and for providing input into efficacy assessments.
* For double blind only: Meet the decline criteria of functional (as assessed by the investigator) and cognitive (assessed by a 1 point reduction in Mini-Mental State Examination) score between visits or a 3 point reduction from baseline) decline at weeks 23, 36 or 48.

Exclusion Criteria:

* Presence of an advanced, severe, progressive, or unstable disease of any type that could interfere with efficacy and safety assessments or put the patient at particular risk,
* Any medical or neurological condition other than Alzheimers Disease that could explain the patient's dementia,
* A diagnosis of probable or possible vascular dementia,
* A current diagnosis of unsuccessfully-treated depression, or any other mental disorder that may interfere with the evaluation of the patient's response to study medication,
* A history or current diagnosis of cerebrovascular disease (e.g. stroke),
* A current diagnosis of severe or unstable cardiovascular disease (e.g. unstable coronary artery disease).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1584 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (143):
- United States (64):
  - Novartis investigative site, Birmingham, Alabama
  - Novartis investigative site, Gilbert, Arizona
  - Novartis investigative site, Phoenix, Arizona
  - Novartis investigative site, Sun City, Arizona
  - Novartis investigative site, Anaheim, California
  - Novartis investigative site, Carson, California
  - Novartis investigative site, Costa Mesa, California
  - Novartis investigative site, Fullerton, California
  - Novartis investigative site, La Habra, California
  - Novartis investigative site, La Jolla, California
  - Novartis investigative site, National City, California
  - Novartis investigative site, Redlands, California
  - Novartis investigative site, San Francisco, California
  - Novartis investigative site, Fort Collins, Colorado
  - Novartis investigative site, Longmont, Colorado
  - Novartis investigative site, Boca Raton, Florida
  - Novartis investigative site, Bradenton, Florida
  - Novartis investigative site, Deerfield Beach, Florida
  - Novartis investigative site, Delray Beach, Florida
  - Novartis investigative site, Fort Lauderdale, Florida
  - Novartis investigative site, Gainesville, Florida
  - Novartis investigative site, Miami Beach, Florida
  - Novartis investigative site, Pompano Beach, Florida
  - Novartis investigative site, Port Charlotte, Florida
  - Novartis investigative site, Sunrise, Florida
  - Novartis investigative site, West Palm Beach, Florida
  - Novartis investigative site, Atlanta, Georgia
  - Novartis investigative site, Macon, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis investigative site, Chicago, Illinois
  - Novartis investigative site, Springfield, Massachusetts
  - Novartis investigative site, Flint, Michigan
  - Novartis investigative site, Flushing, Michigan
  - Novartis investigative site, Roseville, Michigan
  - Novartis investigative site, Traverse City, Michigan
  - Novartis investigative site, Hattiesburg, Mississippi
  - Novartis investigative site, Ocean Springs, Mississippi
  - Novartis investigative site, Columbia, Missouri
  - Novartis investigative site, St Louis, Missouri
  - Novartis investigative site, Flemington, New Jersey
  - Novartis investigative site, Nutley, New Jersey
  - Novartis investigative site, Somerset, New Jersey
  - Novartis investigative site, Albany, New York
  - Novartis investigative site, Syracuse, New York
  - Novartis investigative site, Greensboro, North Carolina
  - Novartis investigative site, Morganton, North Carolina
  - Novartis investigative site, Winston-Salem, North Carolina
  - Novartis investigative site, Canton, Ohio
  - Novartis investigative site, Columbus, Ohio
  - Novartis investigative site, Corvallis, Oregon
  - Novartis investigative site, Portland, Oregon
  - Novartis investigative site, Beaver, Pennsylvania
  - Novartis investigative site, Erie, Pennsylvania
  - Novartis investigative site, Greensburg, Pennsylvania
  - Novartis investigative site, Pittsburgh, Pennsylvania
  - Novartis investigative site, Beaufort, South Carolina
  - Novartis investigative site, Summerville, South Carolina
  - Novartis investigative site, Brentwood, Tennessee
  - Novartis investigative site, Nashville, Tennessee
  - Novartis investigative site, Dallas, Texas
  - Novartis investigative site, Fort Worth, Texas
  - Novartis investigative site, Irving, Texas
  - Novartis investigative site, Charleston, West Virginia
  - Novartis investigative site, Huntington, West Virginia
- Canada (14):
  - Novartis investigative site, Toronto, Ontario
  - Novartis investigative site, Calgary
  - Novartis investigative site, Edmonton
  - Novartis investigative site, Greenfield Park
  - Novartis investigative site, Halifax
  - Novartis investigative site, London
  - Novartis investigative site, Montreal
  - Novartis investigative site, Ottawa
  - Novartis investigative site, Peterborough
  - Novartis investigative site, Québec
  - Novartis investigative site, Regina
  - Novartis investigative site, Toronto
  - Novartis investigative site, Vancouver
  - Novartis investigative site, Winnipeg
- France (14):
  - Novartis investigative site, Fains-Véel, Alsace Lorraine
  - Novartis investigative site, Dijon, Burgundy
  - Novartis investigative site, Reims, Champagne-Ardenne
  - Novartis investigative site, Bordeaux
  - Novartis investigative site, Bourg-en-Bresse
  - Novartis investigative site, Caen
  - Novartis investigative site, Cherbourg
  - Novartis investigative site, Dijon
  - Novartis investigative site, Limoges
  - Novartis investigative site, Montpellier
  - Novartis investigative site, Nice
  - Novartis investigative site, Paris
  - Novartis investigative site, Rennes
  - Novartis investigative site, Rodez
- Germany (19):
  - Novartis investigative site, Bad Neustadt/Saale
  - Novartis investigative site, Berlin
  - Novartis investigative site, Bonn
  - Novartis investigative site, Burg
  - Novartis investigative site, Cologne
  - Novartis investigative site, Düsseldorf
  - Novartis investigative site, Frankfurt
  - Novartis investigative site, Giessen
  - Novartis investigative site, Krefeld
  - Novartis investigative site, Leipzig
  - Novartis investigative site, Magdeburg
  - Novartis investigative site, Mannheim
  - Novartis investigative site, Marburg
  - Novartis investigative site, München
  - Novartis investigative site, Münster
  - Novartis investigative site, Nuremberg
  - Novartis investigative site, Stralsund
  - Novartis investigative site, Stuttgart
  - Novartis investigative site, Würzburg
- Italy (27):
  - Novartis investigative site, Milan, Milan
  - Novartis investigative site, Ancona
  - Novartis investigative site, Arcugnano
  - Novartis investigative site, Arezzo
  - Novartis investigative site, Bari
  - Novartis investigative site, Bologna
  - Novartis investigative site, Brescia
  - Novartis investigative site, Cagliari
  - Novartis investigative site, Catania
  - Novartis investigative site, Città di Castello
  - Novartis investigative site, Cremona
  - Novartis investigative site, Ferrara
  - Novartis investigative site, Florence
  - Novartis investigative site, Foggia
  - Novartis investigative site, Genova
  - Novartis investigative site, La Spezia
  - Novartis investigative site, Milan
  - Novartis investigative site, Modena
  - Novartis investigative site, Napoli
  - Novartis investigative site, Padua
  - Novartis investigative site, Pavia
  - Novartis investigative site, Perugia
  - Novartis investigative site, Pisa
  - Novartis investigative site, Rho
  - Novartis investigative site, Rome
  - Novartis investigative site, Torino
  - Novartis investigative site, Verona
- Spain (2):
  - Novartis investigative site, Barcelona
  - Novartis investigative site, Palma de Mallorca
- Switzerland (3):
  - Novartis investigative site, Basel
  - Novartis investigative site, Biel
  - Novartis investigative site, Mendrisio

REFERENCES:
- [Derived] Molinuevo JL, Frolich L, Grossberg GT, Galvin JE, Cummings JL, Krahnke T, Strohmaier C. Responder analysis of a randomized comparison of the 13.3 mg/24 h and 9.5 mg/24 h rivastigmine patch. Alzheimers Res Ther. 2015 Mar 8;7(1):9. doi: 10.1186/s13195-014-0088-8. eCollection 2015. PMID 25755685
- [Derived] Grossberg G, Cummings J, Frolich L, Bellelli G, Molinuevo JL, Krahnke T, Strohmaier C. Efficacy of higher dose 13.3 mg/24 h rivastigmine patch on instrumental activities of daily living in patients with mild-to-moderate Alzheimer's disease. Am J Alzheimers Dis Other Demen. 2013 Sep;28(6):583-91. doi: 10.1177/1533317513495104. PMID 23982674

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1,584 participants were enrolled, 1582 received study drug during the initial open label period; of these, 567 were qualified to enter a double blind randomized period.
Groups:
- Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2): Rivastigmine 5 cm^2 transdermal patch once a day during the first 4 weeks of open label treatment followed by rivastigmine 10 cm^2 transdermal patch once a day from week 4 to week 24, 36 or 48.
- Extended Open Label (10 cm^2): Rivastigmine 10 cm^2 transdermal patch once a day during 48 weeks (from week 48 to week 96) open label treatment.
Period: Initial Open Label (Maximum 48 Weeks)
Arm/Group | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2) | Extended Open Label (10 cm^2)
Started | 1584 (Enrolled patients.) | 0 | 0 | 0
Exposed to Study Drug | 1582 | 0 | 0 | 0
Completed | 1085 | 0 | 0 | 0
Not Completed | 499 | 0 | 0 | 0
Not completed — Adverse Event | 272 | 0 | 0 | 0
Not completed — Abnormal laboratory value | 1 | 0 | 0 | 0
Not completed — Abnormal test procedure results | 1 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 58 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 88 | 0 | 0 | 0
Not completed — Lost to Follow-up | 22 | 0 | 0 | 0
Not completed — Administrative problem | 7 | 0 | 0 | 0
Not completed — Death | 22 | 0 | 0 | 0
Not completed — Protocol Violation | 28 | 0 | 0 | 0
Period: Double Blind (Maximum 48 Weeks )
Arm/Group | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2) | Extended Open Label (10 cm^2)
Started | 0 | 286 (1 patient was randomized in error and did not receive study drug, hence excluded from this arm.) | 280 | 0
Completed | 0 | 203 | 207 | 0
Not Completed | 0 | 83 | 73 | 0
Not completed — Adverse Event | 0 | 33 | 28 | 0
Not completed — Death | 0 | 5 | 3 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 13 | 13 | 0
Not completed — Protocol Violation | 0 | 5 | 3 | 0
Not completed — Lost to Follow-up | 0 | 4 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 20 | 17 | 0
Not completed — Administrative problems | 0 | 3 | 2 | 0
Not completed — Condition no longer requires study drug | 0 | 0 | 1 | 0
Period: Extended Open Label (Maximum 48 Weeks)
Arm/Group | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2) | Extended Open Label (10 cm^2)
Started | 0 | 0 | 0 | 457 (Two participants did not receive study drug, hence excluded from this arm.)
Completed | 0 | 0 | 0 | 395
Not Completed | 0 | 0 | 0 | 62
Not completed — Administrative problems | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 18
Not completed — Lost to Follow-up | 0 | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 14
Not completed — Protocol Violation | 0 | 0 | 0 | 5
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 6
Not completed — Death | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total Patients: Total number of patients enrolled in the initial open label period that may have been randomized in the double blind period or may have continued in the extended open label period.
Arm/Group | Total Patients
Number analyzed (Participants) | 1584
Age Continuous [Mean (Standard Deviation); unit: years] | 74.93 (7.131)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 992
  Male | 592

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) Subscale at Week 48 of Double Blind Period
Description: The Alzheimer's Disease Assessment Scale-Cognitive (ADAS-cog) subscale comprises 11 items summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment. A negative change indicates an improvement from baseline.
Time Frame: Baseline and week 48 of double blind period
Population: Intent to treat population double blind (ITT-DB): included all randomized patients who received at least 1 dose of double blind study drug, and had at least 1 post-randomization assessment for both co-primary efficacy variables: Alzheimer's Disease Assessment Scale-Cognitive and Disease Cooperative Study-Instrumental Activities of Daily Living.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2)
Number analyzed (Participants) | 268 | 264
units on a scale | 4.9 (7.49) | 4.1 (8.00)

2. Primary Outcome: Change in Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-IADL) Subscale Score From Baseline to Week 48 of Double Blind Period
Description: The Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-IADL) is a 16 item subscale of the caregiver-based ADCS-IADL scale, developed for the use in dementia studies. The ADCS-IADL total score ranges from 0 to 56, with higher scores indicating less severe impairment. A positive change indicates an improvement from baseline.
Time Frame: Baseline and week 48 of double blind period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2)
Number analyzed (Participants) | 271 | 265
units on a scale | -6.2 (8.78) | -4.4 (8.21)

3. Secondary Outcome: Time to Functional Decline as Measured by Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-IADL) Subscale During the Double Blind Period
Description: Functional decline was defined by either an at least 1 point decrease in the Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-IADL) subscale score in a visit and confirmed by the following visit/assessment or at least 2 points decrease from the double blind randomization baseline.
Time Frame: 390 days was the maximum
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Time in days
Arm/Group | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2)
Number analyzed (Participants) | 271 | 265
Time in days | 90 [85 to 113] | 91 [85 to 113]

4. Secondary Outcome: Change in Attention and Executive Function as Assessed by the Trail Making Test (Part A) at Week 48 of the Double Blind Period
Description: Change from baseline to week 48 in total time to perform Trail Making Test (TMT) part A. This test provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. The TMT part A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. The score represents the amount of time required to complete the task. Total values for TMT part A range between 0 and 300 seconds. A negative change indicates an improvement from baseline.
Time Frame: Baseline and week 48 of double blind period
Population: Intent to treat population (ITT-DB): included all randomized patients with an assessment at baseline and week 48 who received at least 1 dose of double blind study drug, and had at least 1 post-randomization assessment for both co-primary efficacy variables (ADAS-cog and ADCS-IADL).
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2)
Number analyzed (Participants) | 258 | 254
Time in seconds | 18.2 (62.57) | 16.3 (66.09)

5. Secondary Outcome: Change in Attention and Executive Function as Assessed by the Trail Making Test (Part B) at Week 48 of Double Blind Period
Description: Change from baseline to week 48 in total time to perform Trail Making Test (TMT) part B. This test provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. TMT has two parts: Part A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-Part B except the person must alternate between numbers and letters. Total values for TMT part B range between 0 and 420 seconds. A negative change from baseline indicates an improvement in condition.
Time Frame: Baseline and week 48 of double blind period
Population: Intent to treat population (ITT-DB): included all randomized patients with an assessment at baseline and week 48 who received at least 1 dose of double blind study drug, and had at least 1 post-randomization assessment for both co-primary efficacy variables (ADAS-cog, ADCS-IADL).
Measure: Mean (Standard Deviation); unit: Time in seconds
Groups:
- Double Blind: Rivastigmine (15 cm^2): Rivastigmine transdermal patch 15 cm^2 and placebo to rivastigmine 10 cm^2 once daily for 48 weeks during the double blind period.
Arm/Group | Double Blind: Rivastigmine (15 cm^2) | Double Blind: Rivastigmine (10 cm^2)
Number analyzed (Participants) | 235 | 236
Time in seconds | 9.3 (68.80) | 5.8 (65.38)

6. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI)-10 Score at Week 48 of Double Blind Period
Description: Change from baseline to week 48 as assessed by the Neuropsychiatric Inventory (NPI)-10 total score. The scale consists of 10 domains that are rated for both frequency (range 1-4) and severity (range 1-3). A composite score for each domain is calculated (frequency x severity) which ranges from 1 to 12. There is a leading question for each item. If the symptom is not present then the frequency, severity and distress scores are not completed. In this case the score is 0 for the item. The sum of the composite scores yields the NPI-10 total score (range 0-120). A negative change in score indicates an improvement from baseline (symptom reduction).
Time Frame: Baseline and week 48 of double blind period
Population: Intent to treat population double blind (ITT-DB): included all randomized patients with an assessment at baseline and week 48, who received at least 1 dose of double blind study drug, and had at least 1 post-randomization assessment for both co-primary efficacy variables (ADAS-cog, ADCS-IADL).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2)
Number analyzed (Participants) | 271 | 265
units on a scale | 0.9 (10.98) | 1.4 (11.51)

7. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Discontinuations Due to Adverse Events
Time Frame: 30 days after a maximum of 96 weeks treatment
Population: The safety set included all patients who received at least one dose of study medication and who had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Groups:
- Double Blind: Rivastigmine (15 cm^2): Rivastigmine transdermal patch 15c m^2 and placebo to rivastigmine 10 cm^2 once daily for 48 weeks during double blind period.
- Extended Open Label (10 cm^2): Rivastigmine 10 cm^2 transdermal patch once a day during 48 weeks open label treatment running in parallel to the double blind period.
Arm/Group | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2) | Extended Open Label (10 cm^2)
Number analyzed (Participants) | 1582 | 283 | 280 | 457
Participants | 1135 | 193 | 210 | 263

ADVERSE EVENTS:
Time Frame: 30 days after a maximum of 96 weeks treatment
Description: The safety set included all patients who received at least one dose of study medication and who had at least one post-baseline safety assessment.
Groups:
- Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2): Safety population Initial Open Label (Safety-IOL) - This population consisted of all patients who received at least 1 dose of study drug during the initial open label phase and had at least 1 post baseline safety assessment during the same phase.
- Double Blind: Rivastigmine (10 cm^2); Double Blind: Rivastigmine (15 cm^2): Safety population Double Blind (Safety-DB) - This population included all patients who were randomized, received at least 1 dose of study drug during the double blind phase and had at least 1 post-randomization safety assessment during the double blind phase. Patients were analyzed according to treatment received.
- Extended Open Label: Rivastigmine (10 cm^2): Safety population Extended Open Label (Safety-EOL) - This population consisted of all patients who received at least 1 dose of study drug during the extended open label phase and had at least 1 post baseline safety assessment during the same phase.
Arm/Group | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) | Double Blind: Rivastigmine (10 cm^2) | Double Blind: Rivastigmine (15 cm^2) | Extended Open Label: Rivastigmine (10 cm^2)
Serious Adverse Events (participants affected / at risk) | 227/1582 | 44/283 | 44/280 | 59/457
Other Adverse Events (participants affected / at risk) | 732/1582 | 110/283 | 151/280 | 112/457
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) (N=1582) | Double Blind: Rivastigmine (10 cm^2) (N=283) | Double Blind: Rivastigmine (15 cm^2) (N=280) | Extended Open Label: Rivastigmine (10 cm^2) (N=457)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 2 | 0 | 1
Aortic valve calcification (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 9 | 2 | 0 | 3
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 3 | 1 | 2 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 8 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 6 | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 2 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 12 | 2 | 3 | 1
Abasia (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Complication of device removal (General disorders) | 0 | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 2
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 2 | 4 | 2
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 4 | 4 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 2 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 12 | 1 | 3 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 7 | 2 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 1
Cardiac enzymes increased (Investigations) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 3 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 1 | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Crying (Nervous system disorders) | 1 | 0 | 0 | 0
Dementia (Nervous system disorders) | 3 | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 3 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 1 | 2 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Multiple system atrophy (Nervous system disorders) | 1 | 0 | 0 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Neurological decompensation (Nervous system disorders) | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 2 | 1
Psychomotor hyperactivity (Nervous system disorders) | 3 | 1 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Senile dementia (Nervous system disorders) | 1 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 14 | 3 | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 3 | 1 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 5 | 2 | 2 | 0
Agitation (Psychiatric disorders) | 6 | 2 | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 4 | 2 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Fear (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 2 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 4 | 1 | 0 | 3
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1 | 2
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 1 | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Open Label: Rivastigmine (5 cm^2 / 10 cm^2) (N=1582) | Double Blind: Rivastigmine (10 cm^2) (N=283) | Double Blind: Rivastigmine (15 cm^2) (N=280) | Extended Open Label: Rivastigmine (10 cm^2) (N=457)
Abdominal pain upper (Gastrointestinal disorders) | 17 | 3 | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 73 | 13 | 18 | 4
Nausea (Gastrointestinal disorders) | 90 | 13 | 33 | 11
Vomiting (Gastrointestinal disorders) | 68 | 12 | 27 | 1
Application site erythema (General disorders) | 184 | 16 | 18 | 10
Application site pruritus (General disorders) | 139 | 11 | 11 | 5
Application site rash (General disorders) | 56 | 5 | 6 | 2
Urinary tract infection (Infections and infestations) | 45 | 8 | 11 | 11
Fall (Injury, poisoning and procedural complications) | 53 | 16 | 19 | 24
Weight decreased (Investigations) | 44 | 8 | 19 | 12
Decreased appetite (Metabolism and nutrition disorders) | 36 | 7 | 16 | 5
Dizziness (Nervous system disorders) | 37 | 2 | 10 | 8
Headache (Nervous system disorders) | 62 | 11 | 11 | 7
Agitation (Psychiatric disorders) | 42 | 14 | 12 | 5
Anxiety (Psychiatric disorders) | 56 | 7 | 10 | 10
Depression (Psychiatric disorders) | 65 | 13 | 14 | 15
Insomnia (Psychiatric disorders) | 40 | 7 | 11 | 6
Urinary incontinence (Renal and urinary disorders) | 25 | 5 | 9 | 6
Hypertension (Vascular disorders) | 53 | 8 | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.